CLINICAL TRIAL: NCT01248598
Title: The Prevelance Rate of Human Cytomegalovirus (HCMV), Epstein-Barr Virus (EBV) and Human Herpes Virus (HHV-6) in a Saliva of the Patient With Periodantitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Department of Periodontology, School of Gradute Dentistry Rambam Health care campus Haifa, Israel
Other Study IDs: 400-10-RMB CTIL
Record Dates: First submitted 2010-11-21; First posted 2010-11-25 (Estimated); Last update posted 2010-11-25 (Estimated); Status verified 2010-10

CONDITIONS: Cytomegalovirus; Epstein-Barr Virus Infections; Herpesvirus Infection
MeSH Terms: conditions — Epstein-Barr Virus Infections; Herpesviridae Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to study the prevalence of EBV, HCMV, HHV-6 in saliva and on the toothbrush patient with periodontitis.

DETAILED DESCRIPTION:
Human cytomegalovirus (HCMV), Epstein-Barr virus (EBV) Human Herpes virus6 (HHV-6)

ELIGIBILITY:
Inclusion Criteria:

* Patient with peridontitis

Exclusion Criteria:

* Previous periodontal treatment in last 3 month
* Toothbrushing disability

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient of the Department of Periodontology, School of Graduate Dentistry Rambam Health care campus
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2010-10

PRIMARY OUTCOMES:
The Prevelance Rate of the EBV, HCMV, HHV-6 in saliva | 1 year
  Check the EBV, HCMV, HHV-6 in saliva by PCR

SECONDARY OUTCOMES:
change outcomes EBV, HCMV, HHV-6 in saliva before and after toothbrushing | 1 year
  Check the EBV, HCMV, HHV-6 in saliva by RC-PCR before and after toothbrushing

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Periodontology, School of Graduate Dentistry Rambam Health care campus, Haifa, Israel